CLINICAL TRIAL: NCT06802068
Title: A Randomized Controlled Clinical Trial Assessing the Impact of 14-week Natural Salmon Oil Supplementation (CARDIO®) on the Omega-3 Index Response and Cardiometabolic and Inflammatory Biomarkers in Healthy, Non-Pregnant Adults
Brief Title: Change in Omega 3 Index in Healthy Adults With OmeGo or a Standard Omega-3 Oil Supplement
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hofseth Biocare ASA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HBC-CARDIO-2024-001-v2
Record Dates: First submitted 2025-01-27; First posted 2025-01-30 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Supplementation in Healthy Adults to Assess Impact on Omega 3 Index and Cardiometabolic Health
Keywords: Omega-3 index, salmon oil CARDIO, omega-3 oil
MeSH Terms: interventions — Cod Liver Oil

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either a whole salmon oil supplement or a cod liver oil supplement.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CARDIO salmon oil soft gel capsules (Active Comparator): A minimally processed, whole salmon oil containing all the fatty acid fractions found in salmon
  Interventions: Dietary Supplement: whole salmon oil
- Omega-3 cod liver oil soft gel capsules (Active Comparator): A standard, processed, concentrated omega-3 supplement
  Interventions: Dietary Supplement: Cod liver oil

INTERVENTIONS:
Dietary Supplement: whole salmon oil — A minimally processed whole salmon oil
  Other Names: CARDIO oil
  Arms: CARDIO salmon oil soft gel capsules
Dietary Supplement: Cod liver oil — Standard, processed omega-3 cod liver oil
  Arms: Omega-3 cod liver oil soft gel capsules

SUMMARY:
Omega-3 index is used as a proxy for an adequate intake of fish unsaturated fats in the diet. However, omega-3 supplements have not consistently shown the health benefits of eating fresh fish. This study will assess the change in omega-3 index and impact on markers of cardiometabolic health with two different supplements: a whole, unprocessed salmon oil and a standard, processed, concentrated oemga-3 oil. The markers to be studies included impact on inflammation and oxidative stress, cholesterol and markers of risk of diabetes. Change in sleep metrics will also be assessed.

DETAILED DESCRIPTION:
Omega-3 index is used as a proxy for an adequate intake of fish unsaturated fats in the diet. However, omega-3 supplements have not consistently shown the health benefits akin to eating fresh fish. This could be because contains many more fats than just EPA and DHA and these other fats have well defined health benefits such as oleic acid which is also abundant in olive oil. Alternatively this might be a result of significant processing needed to extract and concentrate the omega-3 fraction resulting in elevated levels of oxidation and free fatty acids, both of which are pro-inflammatory and would therefore impair the health benefits of omega-3. This study will assess the change in omega-3 index and impact on markers of cardiometabolic health with two different supplements: a whole, unprocessed salmon oil and a standard, processed, concentrated oemga-3 oil. The markers to be studies included impact on common drivers of inflammation and oxidative stress, blood cholesterol and markers of the risk of developing diabetes. Change in sleep metrics will also be assessed using both questionnaires and data from the hypnograms recorded by wearable device.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-pregnant adults; 40-80 years of age; stable body weight prior 3 months

Exclusion Criteria:

* Fish or seafood allergies; Pregnant; already consuming fish oil supplementation; malabsorption states; malignancy in remission for less than 12 months; diabetic

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2025-12-23 (Actual); Study Completion 2026-01-05 (Estimated)

PRIMARY OUTCOMES:
To assess and compare the bioavailability of a natural salmon oil with that of a standard omega-3 supplement | 18 weeks
  Change in omega-3 index after 14 weeks supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Crawford Currie, MBBS, Principal Investigator — HBC
Locations (2):
- United States (2):
  - Alethios, Menlo Park, California
  - Alethios, Inc., San Francisco, California

IPD SHARING:
Plan to Share IPD: Yes
We will put the anonymized data from the study onto the Figshare platform so that journal reviewers and editors can review it as well as other researchers.

REFERENCES:
- [Background] GBD 2017 Diet Collaborators. Health effects of dietary risks in 195 countries, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2019 May 11;393(10184):1958-1972. doi: 10.1016/S0140-6736(19)30041-8. Epub 2019 Apr 4. PMID 30954305